CLINICAL TRIAL: NCT05113095
Title: Postmarketing Surveillance Registry to Evaluate Safety and Efficacy of Darvadstrocel for the Treatment of Complex Perianal Fistulas in Crohn's Disease Patients (J-INSPIRE) (All-case Surveillance)
Brief Title: A Survey of Darvadstrocel in People With Crohn's Disease
Acronym: J-INSPIRE
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Alofisel-5008; jRCT2033210424 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-11-05; First posted 2021-11-09 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Darvadstrocel: Darvadstrocel, 24 mL suspension of 120 million cells as a perilesional injection, once. Participants received interventions as part of routine medical care.
  Interventions: Biological: Darvadstrocel

INTERVENTIONS:
Biological: Darvadstrocel — Darvadstrocel injection
  Other Names: Cx601

SUMMARY:
This study is a survey in Japan of Darvadstrocel injection used to treat Crohn's disease people with complicated anal fistula. The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

The main aim of the study is to check for side effects related from Darvadstrocel injection and to check if Darvadstrocel injection improves symptoms of Crohn's disease. During the study, participants with Crohn's disease will take Darvadstrocel injection according to their clinic's standard practice. The study doctors will check for side effects from Darvadstrocel for 36 months.

ELIGIBILITY:
Inclusion Criteria All patients with complex perianal fistulas in Crohn's Disease who received Darvadstrocel will be included.

Exclusion Criteria None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with complex perianal fistulas in Crohn's Disease who received Darvadstrocel will be included.
Sampling Method: Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 36 Months
  An adverse event is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product. It does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a pharmaceutical product (including an investigational product for a new indication in Japan), whether or not related to the pharmaceutical product.
Percentage of Participants who Achieve Clinical Response | Baseline, Up to Months 36
  Clinical Response is defined as the clinically confirmed closure of at least 50% of the fistulas with this product as compared to baseline that were not drained with gentle finger compression.
Percentage of Participants who Achieve Clinical Remission | Baseline, Up to Months 36
  Clinical remission is defined as the clinically confirmed closure of all fistulas treated with this product as compared to baseline with no discharge despite gentle finger compression.
Percentage of Participants who Achieve Combined Remission | Baseline, Up to Months 36
  Combined remission is defined as the clinically confirmed closure of all baseline external openings that were not drained by gentle finger compression with this product treatment, and absence of an abscess greater than or equal to 2 cm in size confirmed by pelvic MRI (if performed) performed within 6 months of this product treatment.

SECONDARY OUTCOMES:
Percentage of Participants who Occurred Recurrence of Previously Treated Anal Fistulas in Participants who Achieved Clinical Remission at the Previous Visit | Baseline, Up to Months 36
  Recurrence of previously treated anal fistulas in patients who achieved clinical remission at the previous visit is defined as clinically confirmed recurrence with expulsion in any of the external openings treated with this product or the presence of a 2-axis or larger abscess > 2 cm in a previously treated fistula confirmed by MRI scan (if performed).
Percentage of Participants with New Perianal Abscess in a Previously Treated Anal Fistula | Baseline, Up to Months 36
  New perianal abscess in a previously treated anal fistula is defined as fluid collection with a margin enhancing effect such that a high signal on T2-weighted image and a high signal edge on Gadolinium-enhanced T1-weighted image of the pelvis at the site of administration of this product, if performed. A new perianal abscess will be reported as an adverse event and the investigator will determine the causality with this product treatment.
Change from Baseline in Perianal Disease Activity Index (PDAI) | Baseline, Up to Months 36
  The PDAI is a scoring system to evaluate the severity of perianal lesion associated with Crohn's disease. It includes the following 5 items: (a) Discharge; (b) Pain; (c) Restriction of sexual activity; (d) Type of perianal disease; and (e) Degree of induration. The discharge item is graded on a 5-point scale where 0 indicates no symptoms and 4 indicates severe symptoms and total range of score is from 0 to 4. Higher score means more severe disease. Negative change from Baseline indicates improvement.
Change from Baseline in Harvey Bradshaw Index (HBI: Simple CDAI Score) | Baseline, Up to Months 36
  The HBI is a physician-reported index consisting of five clinical manifestations of CD. HBI items include performance status, abdominal pain, number of watery stools per day, abdominal mass, and complications. The HBI is a cumulative scoring system with the following threshold for lesion activity: Remission (< 5), mild (5 ~ 7), moderate (8 ~ 16), severe (> 16). Higher score means more severe disease. Negative change from Baseline indicates improvement.
Health-Related Quality of Life (HRQOL) Measured by EuroQoL Five Dimensions Five Levels (EQ-5D-5L) Scale | Baseline, Up to Months 36
  EQ-5D-5L is a self-administered preference-based measure of health status suitable for calculating quality-adjusted life-years (QALYs) to inform economic evaluations. EQ-5D-5L includes 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and 5 response levels for each domain (no problems, slight problems, moderate problems, severe problems, and extreme problems). Scores ranges from best (100) to worst (0).
HRQOL Measured by Crohn's Anal Fistula Quality of Life (CAF-QoL) Scale | Baseline, Up to Months 36
  CAF-QoL scale is a measure to check QOL related to Crohn's anal fistula. CAF-QoL scale includes 28-item questionnaires in 3 categories (symptoms of anal fistula, influence of treatment for anal fistula, and quality of life), and 5 response levels for each domain and each score (Not at all: 0, Rarely applicable: 1, Neither: 2, Almost Applicable: 3, Very Much Applicable: 4) for 27-item questionnaires and text format for remaining 1 questionnaire. Scores ranges from best (0) to worst (104).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda selected site, Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/61a905f5f571d4002a64b449